CLINICAL TRIAL: NCT06505187
Title: Celecoxib Pain Management Following Superficial Parotidectomy: Opioid Sparing Protocol
Brief Title: Celecoxib for ENT Pain Management
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2023-1527; A539770 (Other: UW- Madison); Protocol Version 7/5/24 (Other: UW- Madison)
Record Dates: First submitted 2024-07-10; First posted 2024-07-17 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-12

CONDITIONS: Parotidectomy
MeSH Terms: interventions — Celecoxib; Acetaminophen; Oxycodone

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Celecoxib for pain management (Experimental): Participants receive celecoxib in addition to Tylenol and oxycodone
  Interventions: Drug: Celecoxib; Drug: Tylenol; Drug: Oxycodone
- Placebo for pain management (Sham Comparator): Participants receive placebo in addition to Tylenol and oxycodone
  Interventions: Drug: Tylenol; Drug: Oxycodone; Drug: placebo

INTERVENTIONS:
Drug: Celecoxib — 200mg every 12 hours
  Arms: Celecoxib for pain management
Drug: Tylenol — 650mg q6h
Drug: Oxycodone — 5mg every 6 hours as needed
Drug: placebo — every 12 hours
  Arms: Placebo for pain management

SUMMARY:
The goal of this clinical trial is to find out whether pain can be managed after an operation with celecoxib instead of oxycodone. The main question it aims to answer is if use of celecoxib plus Tylenol reduces the need for oxycodone.

Researchers will compare the combination of celecoxib and Tylenol to a placebo to find out whether celecoxib works to manage pain.

Participants will:

* Take celecoxib, or a placebo, plus Tylenol with opioids as needed
* Keep a diary of their pain between visits
* Complete questionnaires

DETAILED DESCRIPTION:
Surgeons have a unique opportunity to reduce opioid prescriptions - and therefore potential opioid dependence, morbidity and mortality - by altering prescribing patterns in the perioperative period. This study aims to determine if celecoxib is a viable alternative for acute pain control in the postoperative setting for head and neck surgeries which could significantly reduce the amount of narcotic pain pills in circulation and can be extrapolated to other otolaryngologic procedures.

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand and the willingness to sign a written informed consent document
* Willing to comply with all study procedures and be available for the duration of the study
* Ability to take oral medication
* Undergoing superficial parotidectomy
* Individuals at least 18 years of age
* Adequate organ function as indicated by standard laboratory tests: hematology (complete blood count), clinical chemistry

Exclusion Criteria:

* History of NSAIDs contraindication (severe congestive heart failure, CABG within 14 days, arrhythmias, significant coronary artery disease, cardiomyopathy, severe hepatic impairment, history of peptic ulcer disease or GI bleeding, use of anticoagulation (other than prophylactic aspirin)
* History of uncontrolled hypertension, cerebrovascular accident, sulfa allergy, allergy to celecoxib
* Concurrent use of CYP2C9 potentiator/inhibitor
* Use of investigational drugs, biologics, or devices within 30 days prior to randomization.
* Individuals who are pregnant, lactating or planning on becoming pregnant during the study.
* Not suitable for study participation due to other reasons at the discretion of the investigators.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2025-02-28 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Number of oxycodone pills taken | 7 days
  Total number of oxycodone pills taken during the first 7 days post-operative

SECONDARY OUTCOMES:
Change in pain scores | Baseline (post-operative) to 7 days
  Numerical pain scores will be measured using a post-operative modified brief pain inventory. Participants will rate their pain on a scale of 0-10, where 0 = no pain and 10 = worst pain.
Side effects from medications | 7 days
  Participants will self-report any side effects experienced from medications for the first 7 days post-operative
Drain duration | 7 days
  Length of time participant retains the post-operative drain
Number of post-operative complications | 7 days
  Participants will report any post-operative complications experienced during the first 7 days post-operative

CONTACTS AND LOCATIONS:
Overall Officials: Tiffany Glazer, MD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No